CLINICAL TRIAL: NCT07215221
Title: Implementation of the Novel TBI-RECOVER Intervention in Substance Use Treatment: A Hybrid Type 2 Effectiveness-Implementation Pilot Trial
Brief Title: Implementation of TBI-RECOVER in Substance Use Treatment
Acronym: TBI-RECOVER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kathryn Hyzak, Assistant Professor, Ohio State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20251658; 1K01DA060881-01A1 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury; Substance Use Disorder (SUD)
Keywords: hybrid type 2 effectiveness-implementation; traumatic brain injury; RE-AIM; organizational theory; implementation strategies; implementation mechanisms; substance use disorder treatment; hybrid type 2 trial; cognitive impairment; treatment mechanisms; outpatient substance use treatment
MeSH Terms: conditions — Brain Injuries, Traumatic; Substance-Related Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The study will use a quasi-experimental design with a control and treatment group recruited at separate phases of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TBI-RECOVER treatment arm (Experimental): Patients the treatment arm will be screened for brain injury, and those with a positive screen will receive the full TBI-RECOVER intervention model.
  Interventions: Behavioral: TBI-RECOVER
- Control arm (Active Comparator): Patients in the control arm will be screened for brain injury, and those with a positive screen will receive a brief information and educational sheet.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: TBI-RECOVER — The TBI-RECOVER intervention model consists of three components: 1) a web-based brain injury and cognitive impairment screener using the Online Brain Injury Screening and Support System (OBISSS) of the National Association of State Head Injury Administrators, 2) brief education and information on traumatic brain injury and substance use disorders, and 3) neurocognitive accommodations, or compensatory strategies, for neurological impairment.
  Other Names: Neurologic Informed Care
  Arms: TBI-RECOVER treatment arm
Behavioral: Control — The control condition includes a brief information and educational sheet on traumatic brain injury and substance use disorder, how these two conditions are connected with each other, and a list of suggested accommodations they can use in treatment.
  Arms: Control arm

SUMMARY:
The goal of this hybrid type 2 pilot trial is to understand the implementation and effectiveness of the TBI-RECOVER intervention model (e.g., brain injury screening, cognitive and behavioral challenges screening, and neurocognitive accommodations) on patient retention in outpatient substance use disorder treatment. We will evaluate whether an implementation strategy bundle (e.g., training/education, champions, audit & feedback, facilitation) improves provider use and sustainability of the TBI-RECOVER intervention, and also whether the TBI-RECOVER intervention improves patient symptoms and treatment retention.

ELIGIBILITY:
Patient Inclusion Criteria:

* English-speaking; diagnosed with a substance use disorder; assigned to an outpatient provider for psychotherapy at the treatment clinic participating in the study.

Patient Exclusion Criteria:

* None

Provider Inclusion Criteria:

- All providers employed in the outpatient treatment clinic who deliver psychotherapy are eligible (e.g., social workers, counselors, psychologists).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment retention | 1 year
  The proportion of treatment sessions attended over one year.
BASIS-24 scores | 1 year
  The Behavior and Symptom Identification Scale (BASIS-24) measures six domains: (1) substance use, (2) impulsive/addictive behaviors, (3) relationships with self and others, (4) depression/anxiety, (5) daily living/role functioning, and (6) psychosis. Each item is rated on a 5-point Likert scale, where 0 = lowest symptom severity and 4 = highest symptom severity. Subscales and the overall score are summed and then divided by the number of non-missing items for a total score. There are no clinical cut-offs.

SECONDARY OUTCOMES:
Patient self-efficacy | 9 weeks
  The General Self-Efficacy Scale (GSES) will be used to measure self-efficacy. GSES is a 10-item measure of self-efficacy used in research for patients in treatment for SUDs. Items are measured on a 4-point Likert scale, where 1 = "Not at all true" and 4 = "Exactly true." Items are summed for a total score, with higher scores equating to greater self-efficacy. GSES has strong psychometric properties (α = .76 - .90). GSES will be measured at baseline (after informed consent), 3, 6, and 9 weeks.
Cognitive engagement in treatment | 9 weeks
  We will use the Patient Expectation Questionnaire (CEQ), as well as single-item questions. CEQ is a 6-item questionnaire, with items measured on a 1 to 9, where 1 = "not at all logical" and 9 = "very logical." Questions 4 and 6 are rated on a 0-100% scale. Higher scores equal higher cognitive engagement. We will also ask the following single-item questions to measure cognitive engagement: "I understand the goals of my treatment;" "My therapists' approach to providing care will help me reach my goals." Cognitive engagement will be measured at baseline (after informed consent), 3, 6, and 9 weeks.
Satisfaction with treatment | 9 weeks
  We will use the Treatment Perceptions Questionnaire (TPQ),(52) a 10-item measure of treatment satisfaction. Items measured on a 5-point Likert scale, where higher sum scores equal greater satisfaction with treatment. TPQ will be measured once at 9 weeks.

OTHER OUTCOMES:
Adoption | Up to 4 years
  A provider-level measure of the number and proportion of providers who consent to participation relative to the total number of providers eligible.
Reach | Up to 4 years.
  We define and measure "Reach" using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework. As specified in this framework, "Reach" is an implementation outcome measured as the percentage of patients who received the intervention. Therefore, we will identify patients who received the intervention using the electronic health record and the brain injury screening tool (OBISSS) used for this study. The monthly program census (the denominator for determining the percentage for this measure) will be pulled using the electronic health record. Using these data, proportions of patients who received the intervention each month will be calculated and used to measure "Reach."
Implementation adherence using the Fidelity Verification Review Process | 1 year
  The Fidelity Verification Review Process (FVRP) is a provider-level measure of adherence to implementation of each intervention component, and measured on a 4-point Likert scale, where 1 = "Excellent implementation," 2 = "Strong/sufficient implementation," 3 = "Improvement needed implementation," and 4 = "Serious implementation concerns."
Maintenance | At 6-months during the Sustainment Phase
  The Normalization Measure Development Questionnaire (NoMAD) will be used to measure maintenance of TBI-RECOVER implementation. NoMAD is a a program-level measure with 23-items assessing the level of familiarity, normalization, and utilization of TBI-RECOVER per provider report. Three questions encompass the level of familiarity and use of the intervention on a scale of 0-10, where 0 is "not familiar at all" or "not at all used" and 10 = "Feels completely familiar" or "Completely used/part of work." The remaining 20 questions relate to details of the use of the intervention on a 5-point Likert scale, where 5 = "strongly agree" and 1 = "Strongly disagree." Higher scores equal greater familiarity and maintenance of the intervention. Additional questions allow for the respondent to mark that the question is not relevant to their role, stage of implementation, or intervention."

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlie results in publications.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All de-identified data will be shared as soon as possible, and no later than the time of an associated publication or end of the performance period, whichever comes first. The study data will be stored in the repository for at least 5 years.
Access Criteria: The study metadata and datasets will be submitted to ICPSR. Data will be findable and identifiable through a search of the name of the project PI (Dr. Kathryn Hyzak), project title, or key words associated with the study.